CLINICAL TRIAL: NCT04089813
Title: Effect of Metformin on Chronic Pain After Thoracic Surgery in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Principal Investigator, Xuzhou Medical University
Other Study IDs: XYFY2019-0003
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Chronic Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metformin: Patients use metformin to control blood sugar
  Interventions: Drug: Metformin
- Insulin: Patients use Insulin to control blood sugar

INTERVENTIONS:
Drug: Metformin — Patients use metformin to control blood sugar
  Groups: Metformin

SUMMARY:
Metformin has been found to have more and more functions as a commonly used hypoglycemic drug in clinic. It has been found that metformin has anti-inflammatory, anti-tumor and lipid metabolism regulating effects. Basic studies have shown that metformin as an adjuvant drug combined with gabapentin and tramadol is safe and effective in patients with neuropathic pain. Postoperative chronic pain as a common complication has seriously affected the quality of life and mood of patients after surgery.Some studies have shown that chronic pain after partial operation manifests as neuropathic pain. The effect of metformin on chronic pain after thoracic surgery in patients with diabetes mellitus was observed in this experiment, which was compared with patients taking insulin to control blood sugar.

DETAILED DESCRIPTION:
The analgesic mechanism of metformin may include the following aspects:(1)Metformin relieves neuropathic pain mainly because it can activate adenosine monophosphate-activated protein kinase (AMPK), which plays a crucial role in pain regulation as an important endogenous kinase controlling energy metabolism.(2)In addition, metformin can also inhibit ERK signaling pathway, further inhibit sodium channel, prevent the development of peripheral sensitization and achieve the effect of relieving neuropathic pain. (3)Metformin has been shown to alleviate bone cancer pain in rats by reducing STAT3 phosphorylation.Clinical research in this field is limited to basic research and ethical requirements are rarely reported at home and abroad. Li Chunye et al. of Jiangsu University designed a clinical trial to compare the efficacy of metformin and gabapentin combined with tramadol on neuropathic pain. The results showed that metformin had a better effect.

The incidence of chronic pain after thoracic surgery is higher. Postoperative chronic pain is a complex pain. The nature and mechanism of chronic pain after thoracic surgery are still controversial. Some studies have shown that some chronic pain after thoracic surgery manifests neuropathic pain, the mechanism may be related to surgical incision, nerve injury caused by trauma and increased pain sensitization. Can metformin alleviate chronic pain after surgery? The research on this aspect is still blank at present.This study was designed as a prospective cohort study to observe whether there was a difference in the incidence of chronic pain after thoracoscopic lobectomy between patients taking metformin and patients injecting insulin to control blood sugar.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70
2. Diabetes history. Use metformin or insulin to control blood sugar
3. The type of operation is selective thoracoscopic lobectomy.

Exclusion Criteria:

1. Newly diagnosed diabetic patients at admission
2. Complication of severe cardiopulmonary diseases
3. Refuse to participate in this experiment
4. Participate in other trials
5. Patients with diabetic complications (including diabetic nephropathy, peripheral neuropathy, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 diabetic patients undergoing elective thoracoscopic lobectomy in the Affiliated Hospital of Xuzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2019-12-09 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain after operation | 3 months after operation
  A VAS score greater than or equal to 3 is defined as the presence of chronic pain after surgery.

SECONDARY OUTCOMES:
VAS score at extubation time, 12 hours and 24 hours after operation | extubation time, 12 hours and 24 hours after operation
  A VAS score greater than or equal to 3 is defined as the presence of pain after surgery.
Neuropathic pain score and incidence at 3 months after operation | 3 months after operation
  Assessment of the presence of neuropathic pain by using self-rating scale
Anxiety and Depression Score | 3 months after operation
  Assessment of Anxiety and Depression in Patients by HAMD Depression Scale
Length of ICU stay | an average of 2 days
  Some patients may need to be transferred to ICU.
Length of hospital stay | an average of 10 days
  Total length of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: JinDong Liu, M.S, Study Director — Afliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data(IPD) will be available when this trial is finished and the article have been published.

REFERENCES:
- [Result] Shiers S, Pradhan G, Mwirigi J, Mejia G, Ahmad A, Kroener S, Price T. Neuropathic Pain Creates an Enduring Prefrontal Cortex Dysfunction Corrected by the Type II Diabetic Drug Metformin But Not by Gabapentin. J Neurosci. 2018 Aug 15;38(33):7337-7350. doi: 10.1523/JNEUROSCI.0713-18.2018. Epub 2018 Jul 20. PMID 30030404
- [Result] Pecikoza UB, Tomic MA, Micov AM, Stepanovic-Petrovic RM. Metformin Synergizes With Conventional and Adjuvant Analgesic Drugs to Reduce Inflammatory Hyperalgesia in Rats. Anesth Analg. 2017 Apr;124(4):1317-1329. doi: 10.1213/ANE.0000000000001561. PMID 27669556
- [Result] Smith B, Ang D. Metformin: Potential analgesic? Pain Med. 2015 Dec;16(12):2256-60. doi: 10.1111/pme.12816. Epub 2015 May 29. PMID 26031427
- [Result] Ge A, Wang S, Miao B, Yan M. Effects of metformin on the expression of AMPK and STAT3 in the spinal dorsal horn of rats with neuropathic pain. Mol Med Rep. 2018 Apr;17(4):5229-5237. doi: 10.3892/mmr.2018.8541. Epub 2018 Feb 1. PMID 29393487